CLINICAL TRIAL: NCT05941299
Title: A Pivotal Study of REGENERA Implant in Malignant Breast Lesion Treated by Lumpectomy
Brief Title: Safety and Performance of REGENERA Breast Implant in Women Affected by Malignant Breast Lesion Treated by Lumpectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tensive SRL (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Tens-BBC/003/2021
Record Dates: First submitted 2023-06-16; First posted 2023-07-12 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Mastectomy, Segmental; Breast Neoplasm Malignant Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- REGENERA breast implant implantation (Experimental): Single monolateral breast implant
  Interventions: Device: REGENERA breast implant implantation

INTERVENTIONS:
Device: REGENERA breast implant implantation — Each patient will perform 13 study visits, and at each visit, all necessary study procedures will be performed according to the clinical investigation plan:
  * Screening
  * Pre-surgery treatment
  * Surgery and study device implant
  * Post-surgery follow-up

SUMMARY:
The goals of this clinical trial are:

* demonstrate the safety of REGENERA breast implant in patients undergoing lumpectomy of malignant breast lesions
* demonstrate the safety and performance of REGENERA in terms of investigator's satisfaction, potential interference with current standard-of-care imaging techniques and occurrence of device-related serious adverse events.

DETAILED DESCRIPTION:
Participants will perform 13 study visits, and at each visit, all necessary study procedures will be performed according to the clinical investigation plan:

* Screening
* Pre-surgery treatment
* Surgery and study device implant
* Post-surgery follow-up up to 5 years

ELIGIBILITY:
Inclusion Criteria:

* Female adult subject aged 40-70 years.
* Subject diagnosed with malignant breast lesion:
* monolateral nodular infiltrative carcinoma,
* without microcalcification,
* single or multifocal,
* included in an area with a maximum diameter of 4 cm,
* non-metastatic (M0).
* Subject with clinically negative axilla.
* Subject considered eligible for conservative breast surgery - BCS (Breast-Conserving Surgery, lumpectomy or quadrantectomy), leaving a volume deficit compatible with a REGENERA implant (available in two dried sizes) volume of 70 ml or 100 ml.
* Confirmation of malignant lesion (pT1, pT2, pN0, pN1) with no discordance between biopsy and radiological imaging.
* Adequate hematopoietic functions.
* Good general health and mentally sound.
* Subject able and willing to give written informed consent form.

Exclusion Criteria:

* Subject with actual concomitant benign breast lesion (B2 and B3), unless present in the same mammary quadrant or in the contralateral breast.
* Subject with actual concomitant malignancies, lobular neoplasm, metastatic breast carcinoma, sarcoma, malignant phyllodes lesions, or Paget's disease.
* Axillary dissection planned as part of the breast lesion surgery.
* History of surgery, chemotherapy, neoadjuvant chemotherapy, or irradiation of the breast parenchyma object of the study.
* Skin retraction at the breast to be operated.
* Infection of the surgical site confirmed pre-operatively by clinical examination.
* Abnormal blood sugar and glycosylated hemoglobin.
* Hard smoker (more than 10 cigarettes a day).
* Acute or chronic severe renal insufficiency (creatinine values >180 μmol/l).
* History of severe asthma or allergies (including allergy to anesthetics or contrast media).
* Autoimmune disease.
* Subjects who are known to be carriers of BCRA mutation.
* Inability to undergo MRI or allergy to contrast media.
* Systemic infections in an active phase.
* Immunocompromised patients (HIV).
* Pregnant or breastfeeding woman or woman who has nursed a child within 3 months prior to enrolment in the study.
* Subject who has participated in another interventional study within the past 3 months.
* Subject who received immunosuppressant therapy in the last 3 months.
* History of substance abuse (drug or alcohol).
* Non-collaborative patients (severe physical disabilities or psychiatric disorders, as per specialist opinion).

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse events (AEs) with a causal relationship to REGENERA at 3 months. | 3 months
  The rate of AEs with a causal relationship to REGENERA should be <5% at 3 months after implant.

SECONDARY OUTCOMES:
Mean investigator's satisfaction on the implanting procedure at 1week. | 1 week after implant
  At least 7 in a 0-10 Visual Analogue Scale, VAS.
Mean investigator's satisfaction on REGENERA usability during surgery at 1 week. | 1 week after implant
  At least 40 in an "ad hoc" questionnaire (12-60 scale).
Mean investigator's satisfaction on overall surgical procedure and clinical outcome of the patient at 12 months. | 12 months
  At least 7 in a 0-10 Visual Analogue Scale, VAS.
Number of interference events of REGENERA with ultrasound imaging technique, through the completion of a questionnaire by the investigators. | After 6 and 12 months
  An imaging evaluation questionnaire will be provided for investigators to fill out.
Number of interference events of REGENERA with mammography imaging technique, through the completion of a questionnaire by the investigators. | After 12 months
  An imaging evaluation questionnaire will be provided for investigators to fill out.
Number of interference events of REGENERA with MRI (with and without contrast) imaging technique, through the completion of a questionnaire by the investigators. | After 6 and 18 months
  An imaging evaluation questionnaire will be provided for investigators to fill out.
Rate of serious adverse events (SAEs) with a causal relationship to REGENERA after 3 months and up to 18 months. | After 3 months and up to 18 months
  The rate of REGENERA-related SAEs should be <5% at each follow-up after 3 months and up to 18 months.
Rate of SAEs with a causal relationship to REGENERA after 18 months and up to 5 years. | After 18 months and up to 5 years
  The rate of REGENERA-related SAEs should be <7% at each follow-up after 18 months and up to 5 years.

CONTACTS AND LOCATIONS:
Locations (3):
- Italy (2):
  - IEO Istituto Europeo di Oncologia, Milan
  - A.O.U. Pisana - Ospedale Santa Chiara, Pisa
- Complejo Hospitalario Universitario A Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lisa AVE, Bottoni M, Ghilli M, Mariniello MD, Intra M, Belloni LM, Mattar D, Cossu MC, Montrone S, Tamplenizza M, Gerges I, Tocchio A, Acea B, Roncella M, Rietjens M. Volume replacement procedure adopting biomaterial: early considerations from a multicentric study. Updates Surg. 2025 Sep;77(5):1665-1671. doi: 10.1007/s13304-025-02212-2. Epub 2025 Apr 28. PMID 40295450